CLINICAL TRIAL: NCT01655433
Title: VELOCITY: Pilot Study to Evaluate Ultrafast Hypothermia Before Reperfusion in Patients With Acute ST-Elevation Myocardial Infarction
Brief Title: Evaluation of Ultrafast Hypothermia Before Reperfusion in STEMI Patients
Acronym: VELOCITY
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor business decision, not safety related
Sponsor: Velomedix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VMXP-2490
Record Dates: First submitted 2012-07-30; First posted 2012-08-01 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-07

CONDITIONS: ST-elevation MI; Hypothermia
Keywords: ST-elevation MI; Hypothermia
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Therapeutic Hypothermia Treatment (Experimental)
  Interventions: Device: Velomedix APLS device
- No Hypothermia Treatment (Active Comparator): control group is no hypothermia treatment
  Interventions: Other: No Hypothermia Treatment

INTERVENTIONS:
Device: Velomedix APLS device — Velomedix, Automated Peritoneal Lavage System
  Arms: Therapeutic Hypothermia Treatment
Other: No Hypothermia Treatment
  Arms: No Hypothermia Treatment

SUMMARY:
This study will look at the safety of treating patients with heart attack with mild hypothermia induced using a system of automated peritoneal lavage. The hypothesis is that the Velomedix Automated Peritoneal Lavage System can treat patients with heart attack safely and with adequate performance.

DETAILED DESCRIPTION:
The study aims to determine the safety and feasibility of using the Velomedix Automated Peritoneal Lavage System to treat patients with STEMI using therapeutic hypothermia. Patients will undergo cooling, maintenance and rewarming and applicable data will be gathered on device performance and patient safety. Patient temperature and vital signs will be monitored in addition to various laboratory values. Adverse event reporting will take place at multiple time intervals and follow-up will continue out to 6-months.

ELIGIBILITY:
Inclusion Criteria:

* Clinical symptoms consistent with acute STEMI lasting at least 30 minutes
* STEMI with ST-Elevation of ≥2 mm in two or more contiguous ECG leads
* Patient eligible for PCI

Exclusion Criteria:

* Cardiac arrest with return of spontaneous circulation
* Known prior history of MI
* Known history of severe COPD requiring supplemental home oxygen
* Patient experiencing intractable cardiogenic shock, or requiring immediate placement of a mechanical cardiac assist device
* Known severe anemia or abnormal platelet count
* Known significant renal insufficiency
* Known contraindication for MRI
* Known contraindications to hypothermia, such as temperature-sensitive hematological dyscrasias or vasospastic disorders

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2012-11; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Composite of new-onset SAEs | 30 days
  Composite of new-onset serious adverse events, specifically death, ischemia driven target vessel revascularization (TVR), recurrent MI, pneumonia, sepsis, ventricular tachycardia or fibrillation requiring cardioversion, renal failure, peritonitis and significant bleeding.

SECONDARY OUTCOMES:
MACE rate | 30 days
  MACE (cardiac related mortality, recurrent MI, or ischemia driven target vessel revascularization (PCI or CABG) at 30 days
All cause mortality | 6 months
  All cause mortality through 6 months
Myocardial infarct size | 3 days
  Myocardial infarct size at 3 days post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Gregg Stone, MD, Principal Investigator — New York Presbyterian Hospital / Columbia University Medical Center; Graham Nichol, MD, Principal Investigator — University of Washington, Harberview Center
Locations (7):
- United States (5):
  - Heart Center Research, LLC, Huntsville, Alabama
  - LA County USC Hospital, Los Angeles, California
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Ochsner Medical Center, New Orleans, Louisiana
  - Vanderbilt University, Nashville, Tennessee
- Canada (2):
  - Victoria Heart Institute Foundation, Victoria, British Columbia
  - Institut Universitaire de cardiologie et pneumologie de Québec (Hopital Laval), Québec, Quebec

REFERENCES:
- [Derived] Nichol G, Strickland W, Shavelle D, Maehara A, Ben-Yehuda O, Genereux P, Dressler O, Parvataneni R, Nichols M, McPherson J, Barbeau G, Laddu A, Elrod JA, Tully GW, Ivanhoe R, Stone GW; VELOCITY Investigators. Prospective, multicenter, randomized, controlled pilot trial of peritoneal hypothermia in patients with ST-segment- elevation myocardial infarction. Circ Cardiovasc Interv. 2015 Mar;8(3):e001965. doi: 10.1161/CIRCINTERVENTIONS.114.001965. Epub 2015 Feb 19. PMID 25699687